CLINICAL TRIAL: NCT00294840
Title: Dynamic FDG-PET in Aggressive Lymphoma and Pancreas Cancer
Brief Title: Dynamic PET acquisition-a Quantitative Technique for Grading of Malignant Tumors and Prediction of Response to Treatment
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr. Alex Frenkel, Rambam HealthCare Campus
Other Study IDs: PETDCTIL
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2008-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

INTERVENTIONS:
Device: PET-CT

SUMMARY:
To assess a quantitative kinetic model of FDG uptake measurement using PET in patients with aggressive Non-Hodgkin's lymphoma and cancer of the pancreas, malignancies with known variability in disease aggressiveness and prognosis, for optimized tailoring of the therapeutic strategy in the individual patient.

ELIGIBILITY:
Inclusion Criteria:

* age>18
* newly diagnosed untreated aggressive NHL
* newly diagnosed untreated cancer of pancreas

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pancreatric cancer
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The impact of the imaging modality on patient management | 5 years

SECONDARY OUTCOMES:
patient management | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Ora Israel, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Medical Center, Haifa, Israel